CLINICAL TRIAL: NCT01018459
Title: A Phase I Randomized, Controlled, Double-Blinded, Dosage-Escalation Trial to Evaluate the Immunogenicity, Safety, and Reactogenicity of an Adenovirus Type 35 Based Circumsporozoite Malaria Vaccine in Burkinabè, Semi-Immune, Healthy Adults 18 to 45 Years of Age
Brief Title: Adenovirus Type 35 Based Circumsporozoite Malaria Vaccine in Burkina Faso
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-0037
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2012-02

CONDITIONS: Malaria
Keywords: malaria, vaccine, Burkina Faso
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Group D: 10^11 vp/mL or placebo (Experimental): 10 subjects will receive 10^11 vp/mL Ad35.CS.01 and 2 subjects will receive placebo at 0, 1 and 3 months.
  Interventions: Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine; Drug: Placebo
- Group A: 10^9 vp/mL or placebo (Experimental): 10 subjects will receive 10^9 viral particles (vp)/mL Ad35.CS.01 and 2 subjects will receive placebo at 0, 1 and 3 months.
  Interventions: Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine; Drug: Placebo
- Group B: 10^10 vp/mL or placebo (Experimental): 10 subjects will receive 10^10 vp/mL Ad35.CS.01 and 2 subjects will receive placebo at 0, 1 and 3 months.
  Interventions: Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine; Drug: Placebo
- Group C: 5 x 10^10 vp/mL or placebo (Experimental): 10 subjects will receive 5 x 10^10 vp/mL Ad35.CS.01 and 2 subjects will receive placebo at 0, 1 and 3 months.
  Interventions: Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine; Drug: Placebo

INTERVENTIONS:
Biological: Ad35.CS.01 Circumsporozoite Malaria Vaccine — Ad35.CS.01 appears clear to slightly opalescent with no visible particles. Each 0.75 mL dose of the assigned dosage will be administered via intramuscular injection into the deltoid muscle. Dosages: 10^9 viral particles (vp)/mL, 10^10 vp/mL, 5 x 10^10 vp/mL, and 10^11 vp/mL.
Drug: Placebo — Normal saline placebo control delivered via intramuscular injection into the deltoid muscle.

SUMMARY:
The purpose of this study is to evaluate the safety of a malaria vaccine, Ad35.CS.01, and how the body reacts to vaccination. Participants will include 48 Berkinabè healthy males and females ages 18-45 years in Burkina Faso. Volunteers for this study will be divided into 4 groups. Members of each group (12 per group) will receive an increasing dose of vaccine or placebo (an inactive substance). Ten will receive the malaria vaccine and 2 will receive placebo. Study procedures include: physical exam, urine sample, and blood samples. Participants will be involved in study related procedures for about 13 months.

DETAILED DESCRIPTION:
Malaria currently represents one of the most prevalent infections in tropical and subtropical areas throughout the world. Each year, malaria affects around 300 million people and kills 1 to 3 million people in developing countries. Malaria is caused by the mosquito-borne hematoprotozoan parasites belonging to the genus Plasmodium (P.). Malaria parasites have a life cycle consisting of several stages. Each one of these stages is able to induce specific immune responses against the corresponding stage-specific antigens. Malaria parasites are transmitted to man by several species of female Anopheles mosquitoes. Infected mosquitoes inject the sporozoite form of the malaria parasite into the mammalian bloodstream. Before invading hepatocytes, sporozoites remain for a few minutes in the circulation. At this stage the parasite is located in the extracellular environment and is exposed to antibody attack, mainly directed to the circumsporozoite (CS) protein, a major component of the sporozoite surface. Once in the liver, the parasites replicate and develop into schizonts (up to 20,000 per infected cell). During this intracellular stage of the parasite, the main effectors of the host immune response are T lymphocytes, especially CD8+ T cells. Ad35.CS.01 is a malaria vaccine for which a codon optimized nucleotide sequence representing the P. falciparum circumsporozoite (CS) surface antigen is inserted in a replication deficient Adenovirus 35 backbone. It is hypothesized that the Ad35.CS.01 vaccine will prevent the P. falciparum parasite, which causes malaria, from entering and developing within the liver of those who become infected. Ad35.CS.01 would therefore be expected to reduce malaria-attributable morbidity and mortality. The primary objective is to assess the safety and reactogenicity of 4 ascending dosages of Adenovirus Type 35 circumsporozoite malaria vaccine among healthy, semi-immune, subjects given in 3 doses at 0, 1 and 3 months by intramuscular (IM) injection. The secondary objective is to evaluate the immunogenicity of the Adenovirus Type 35 based circumsporozoite malaria vaccine through performance of Humoral Immune Assays (ELISA [enzyme-linked immunosorbent assay] for antibodies to circumsporozoite antigen and Adenovirus Neutralization Assay for neutralizing antibodies to Adenovirus Type 35) and Cellular Immune Assays (Elispot and Flow Cytometry) for CS-specific CD4+ and CD8+ T cell responses and a whole blood ELISA assay to measure secreted cytokines. This is a phase I randomized, controlled, double-blinded, dosage-escalation trial to evaluate the immunogenicity, safety, and reactogenicity of an Adenovirus Type 35 based circumsporozoite malaria vaccine in Burkinabè, in semi-immune, healthy adults 18 to 45 years of age. Researchers propose to confirm the safety of each dosage of the new vaccine by assessing safety laboratory parameters and reactogenicity for 14 days after the initial dose in the lower dosages before escalating to the next dosage level. Each dosage level group will include 10 subjects given vaccine intramuscularly. Two subjects in each dosage group will receive normal saline as placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before any protocol procedures are performed.
* Males and non-pregnant, non-lactating females between the ages of 18 and 45 years, inclusive.
* Females and males must agree to practice adequate contraception until at least 28 days following their last immunization dose (including abstinence; hormonal contraception; condoms with spermicidal agents; post-menopausal; or surgical sterilization/vasectomy).
* Participants must agree to avoid high risk sexual behavior for exposure to human immunodeficiency virus (HIV).
* In good health as determined by screening medical history, physical examination (PE), and laboratory assessments.
* Willingness to comply with protocol requirements.
* Willingness to be contacted for one year for assessment of serious adverse events.
* Must be a permanent resident of the Saponé health district (villages around Balonghin) in Burkina Faso.

Exclusion Criteria:

* Current or recent (within the last four weeks) treatment with parenteral, inhaled, or oral corticosteroids (intranasal steroids are acceptable), or other immunosuppressive agents, or chemotherapy.
* History of splenectomy.
* Abnormal screening laboratory values. Any abnormal screening value for any screening test will exclude the subject from the study. Abnormal screening labs will not be repeated with the exception of high glucose levels will be repeated at a fasting state.
* History of intravenous (IV) drug abuse.
* History of, or current medical, occupational, social or family problems as a result of alcohol or illicit drug use.
* History of moderate to severe mental illness, as defined by symptoms interfering with social or occupational function or suicidal thoughts/attempts.
* History of receiving blood or blood products (such as blood transfusion, platelet transfusion, immunoglobulins, hyperimmune serum) in the previous 6 months.
* Vaccination with a live vaccine within the past 30 days or with a nonreplicating, inactivated, or subunit vaccine within the last 14 days.
* Known hypersensitivity to components of the vaccine.
* History of acute or chronic medical conditions including, but not limited to, disorders of the liver, kidney, lung, heart, or nervous system, or other metabolic or autoimmune/inflammatory conditions.
* History of coagulation defect or bleeding from (bruising at) multiple sites that cannot be linked to trauma or surgery.
* History of anaphylaxis or severe hypersensitivity reaction.
* Severe asthma, as defined by an emergency room visit or hospitalization within the last 12 months.
* Pregnant or breastfeeding women.
* Acute illness, including temperature >37.8 degrees Celsius within one week prior to vaccination.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg).
* Concurrent participation in other investigational protocols or receipt of an investigational product within the previous 30 days or planned receipt of an investigational product within 28 days following the last immunization dose.
* Identification of any condition that, in the opinion of the investigator, would affect the ability of the subject to understand or comply with the study protocol or would jeopardize the safety or rights of a subject participating in the study.
* History of malignancy, including hematologic and skin cancers (except for a localized basal cell carcinoma), or known immunodeficiency syndrome.
* History of previous receipt of a malaria vaccine.
* Pre-medication with analgesic or antipyretic agents in the 6 hours prior to vaccination, or planned medication with analgesic or antipyretic in the 24 hours following vaccination. This criterion should not preclude subjects receiving such medication if the need arises.
* Receipt of a recombinant adenovirus vector vaccine in a prior study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing severe (Grade 3) solicited injection site reactions. | Within 14 days following vaccination.
The number of subjects spontaneously reporting severe (Grade 3) adverse events considered associated with the vaccination. | At any point during the study period.
The number of subjects experiencing severe (Grade 3) solicited systemic reactions | Within 14 days following vaccination.
Serious adverse events considered associated with the vaccination reported. | At any point during the study period.

SECONDARY OUTCOMES:
Neutralizing antibody titers against Adenovirus type 35 by Adenovirus Neutralization Assay. | At days 0, 28, 56, 84, 112 and 140.
Antibody titers against the malaria circumsporozoite antigen [Geometric Mean Titer and individual log enzyme-linked immunosorbent assay (ELISA) units]. | At days 0, 28, 56, 84, 112 and 140.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre National de Recherche et de Formation sur le Paludisme - Research and Training, West Africa, Burkina Faso

REFERENCES:
- [Result] Ouedraogo A, Tiono AB, Kargougou D, Yaro JB, Ouedraogo E, Kabore Y, Kangoye D, Bougouma EC, Gansane A, Henri N, Diarra A, Sanon S, Soulama I, Konate AT, Watson NL, Brown V, Hendriks J, Pau MG, Versteege I, Wiesken E, Sadoff J, Nebie I, Sirima SB. A phase 1b randomized, controlled, double-blinded dosage-escalation trial to evaluate the safety, reactogenicity and immunogenicity of an adenovirus type 35 based circumsporozoite malaria vaccine in Burkinabe healthy adults 18 to 45 years of age. PLoS One. 2013 Nov 11;8(11):e78679. doi: 10.1371/journal.pone.0078679. eCollection 2013. PMID 24244339